CLINICAL TRIAL: NCT05577000
Title: A Phase 1b Clinical Trial of Anti-BCMA Chimeric Antigen Receptor T Cells for Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: Anti-BCMA Chimeric Antigen Receptor T Cells for Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Martin, MD (Other)
Collaborators: Actavis Inc. (Industry); University of California, Davis (Other); Eugia Pharma Specialities Limited (Unknown)
Responsible Party: Sponsor-Investigator, Thomas Martin, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22702; NCI-2022-08957 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-10-08; First posted 2022-10-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Refractory Multiple Myeloma; Relapsed Multiple Myeloma
Keywords: CAR-T Therapies
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (150 x 10^6 CAR + T cells/ infusion) (Experimental): Participants will undergo apheresis with collection of autologous peripheral blood mononuclear cells that will be used to generate CAR-T cells. After successful generation of the anti-BCMA CAR-T cells, participants will undergo lymphodepleting chemotherapy with fludarabine and cyclophosphamide followed by 2-5 days of rest. A single infusion of anti-BCMA CAR-T cells at the starting dose of 150 x 10^6 flat dose will then be given on Day 1.
  Interventions: Biological: Manufactured Anti-BCMA CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Escalation (450 x 10^6 CAR + T cells/ infusion) (Experimental): Participants will undergo apheresis with collection of autologous peripheral blood mononuclear cells that will be used to generate CAR-T cells. After successful generation of the anti-BCMA CAR-T cells, and no dose limiting toxicities were reported for the previous dose level, participants will undergo lymphodepleting chemotherapy with fludarabine and cyclophosphamide followed by 2-5 days of rest. A single infusion of anti-BCMA CAR-T cells at the next highest dose of 450 x 10^6 flat dose will then be given on Day 1.
  Interventions: Biological: Manufactured Anti-BCMA CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Escalation (600 x 10^6 CAR + T cells/ infusion) (Experimental): Participants will undergo apheresis with collection of autologous peripheral blood mononuclear cells that will be used to generate CAR-T cells. After successful generation of the anti-BCMA CAR-T cells, and no dose limiting toxicities were reported for the previous dose level, participants will undergo lymphodepleting chemotherapy with fludarabine and cyclophosphamide followed by 2-5 days of rest. A single infusion of anti-BCMA CAR-T cells at the next highest dose of 600 x 10^6 flat dose will then be given on Day 1.
  Interventions: Biological: Manufactured Anti-BCMA CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Expansion: Maximum Tolerated Dose (MTD) (Experimental): Participants will undergo apheresis with collection of autologous peripheral blood mononuclear cells that will be used to generate CAR-T cells. After successful generation of the anti-BCMA CAR-T cells, and no dose limiting toxicities were reported for the previous dose level, participants will undergo lymphodepleting chemotherapy with fludarabine and cyclophosphamide followed by 2-5 days of rest. A single infusion of anti-BCMA CAR-T cells at the MTD will then be given on Day 1.
  Interventions: Biological: Manufactured Anti-BCMA CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Manufactured Anti-BCMA CAR-T cells — Given IV
  Other Names: Anti-BCMA CAR-T cells
Drug: Fludarabine — Given IV
  Other Names: Fludara
Drug: Cyclophosphamide — Given IV
  Other Names: Cytoxan

SUMMARY:
This is an open-label study to determine the safety of anti-B-cell maturation antigen (BCMA) Chimeric antigen receptor T-cell (CAR T) therapy in participants with Relapsed or Refractory Multiple Myeloma (RRMM).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1. To evaluate the safety of administering chimeric antigen receptor (CAR)-T cells targeting BCMA to participants with RRMM (Dose Escalation).
2. To determine the maximum tolerated dose (MTD) for anti-BCMA CAR-T cells (Dose Escalation).
3. Determine whether administering chimeric antigen receptor T cells targeting BCMA to participants with RRMM increases the overall response rate (ORR) in RRMM compared with historical data for non-CAR agents per International Myeloma Working Group (IMWG) response criteria (Dose Expansion).

SECONDARY OBJECTIVES:

Dose Expansion Only:

1. To describe the efficacy of CAR-T cells targeting BCMA in participants with RRMM.
2. To evaluate the feasibility of manufacturing anti-BCMA CAR-T cells locally and ability to produce adequate quantities of vector positive T-cells.
3. To evaluate the safety and toxicity of CAR-T cells targeting BCMA to participants with RRMM

OUTLINE:

Participants will be enrolled sequentially to each dose level dependent on analysis of dose-limiting toxicities at the previous dose level. A dose expansion will occur at the maximum tolerated dose (MTD). Participants will undergo apheresis with collection of autologous peripheral blood mononuclear cells that will be used to generate CAR-T cells. After successful generation of the anti-BCMA CAR-T cells drug product (DP), participants will undergo lymphodepleting chemotherapy with fludarabine (and cyclophosphamide. Participants will undergo an additional evaluation of eligibility on Day -1 or 1 prior to infusion of anti-BCMA CAR-T cell product. A single infusion of anti-BCMA CAR-T cells at the starting dose will be given on Day 1. Following treatment with DP, participants will be followed up at 12 months and annually for up to 15 years.

ELIGIBILITY:
Eligibility for enrollment:

Inclusion Criteria:

1. Voluntarily sign informed consent form
2. >=18 years of age at the time of signing informed consent
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
4. Diagnosis of MM with relapsed or refractory disease and have had at least 3 different prior lines of therapy including proteasome inhibitor (PI; e.g., bortezomib or carfilzomib) immunomodulatory therapy (IMiD; e.g., lenalidomide or pomalidomide), and anti-CD38 antibody therapy
5. Participants must have measurable disease, including at least one of the criteria below:

   1. Serum M-protein greater or equal to 0.5 g/dL.
   2. Urine M-protein greater or equal to 200 mg/24 h.
   3. Serum free light chain (FLC) assay: involved FLC level of >= 100 mg/L.
6. Adequate organ function, defined as:

   1. Hemoglobulin >8 gm/dl (transfusions allowed).
   2. Platelets >50,000/microliter (uL) (in the absence of platelet transfusion within 7 days of apheresis, but transfusion permitted prior to lymphodepleting chemotherapy).
   3. Absolute neutrophil count (ANC) > 1000/uL in the absence of growth factor support (filgrastim within 7 days or pegfilgrastim within 14 days of apheresis, but growth factor permitted prior to lymphodepleting chemotherapy).
   4. Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 3 x institutional upper limit of normal (ULN).
   5. Total bilirubin =< 1.5 mg/dl x institutional ULN, except with Gilbert's syndrome.
   6. Serum creatinine clearance (CrCl) >= 45 mL/min using Cockcroft-Gault formula.
   7. Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) >= 40% as assessed by echocardiogram or multiple uptake gated acquisition (MUGA).
7. Women of childbearing potential (defined as all women physiologically capable of becoming pregnant) must have a negative serum or urine pregnancy test AND agree to use highly effective methods of contraception for 1 year after the last dose of anti-BCMA CAR-T cells.
8. Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method.

Exclusion Criteria:

1. Autologous transplant within 6 weeks of planned CAR-T cell infusion.
2. Active other malignancy, other than non-melanoma skin cancer, carcinoma in situ (e.g., cervix, bladder, or breast). Any fully treated malignancies or indolent, clinically insignificant malignancies can be discussed among the study team to determine eligibility.
3. HIV seropositivity.
4. Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded).
5. Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, pulmonary abnormalities, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study. NOTE: Women of childbearing potential must have a negative serum or urine pregnancy test.
7. Patients with currently symptomatic central nervous system (CNS) pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia, and Parkinson's disease.
8. History of autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medication within 6 months.

Eligibility for Infusion of Investigational Product:

Includes the inclusion/exclusion criteria required for enrollment with the following exceptions and additions.

Inclusion criteria exceptions:

1. Hematologic function parameters will not be included as a pre-infusion eligibility criterion (because lymphodepletive chemotherapy is expected to cause pancytopenia).
2. Laboratory result abnormalities that are considered not clinically significant by the principal investigator, AND are not the result of a demonstrated active infection or an active central nervous system condition.

Exclusion criteria additions:

1. Use of anti-multiple myeloma therapy, including systemic corticosteroids within 14 days prior to lymphodepletive chemotherapy.
2. Neurologic symptoms suggestive of an active central nervous system condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2043-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events (AE) (Dose Escalation) | From initiation of study treatment (day 1) to 29 days following CAR-T infusion
  Proportion of participants with treatment-emergent adverse events of CAR-T as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0, revised cytokine release syndromeCRS grading criteria (for CRS), and American Society of Transplantation and Cellular Therapy (ASTCT) Immune Effector Cell Associated Neurotoxicity (ICANS) Consensus Grading for Adults (for neurotoxicity).
Proportion of participants who experience a dose-limiting toxicity (DLT) (Dose Escalation) | From initiation of study treatment (day 1) to 29 days following CAR-T infusion
  The DLT evaluable analysis set includes all participants in the dose-finding part of the study who have received the anti-BCMA CAR-T cell product, and who have either experienced a DLT or were followed for the full DLT evaluation period (within 28 days following infusion of CAR-T cells targeting BCMA). The MTD is defined as the dose level immediately below that in which >=2/6 participants experience a DLT and will be used to determine the recommended Phase 2 dose for future studies.
Overall Response Rate (ORR) | Up to 12 months following CAR- T infusion
  Overall response rate includes participants with a demonstrated Stringent Complete Response (sCR), Complete Response (CR), Partial Response (PR), or Very Good Partial Response (VGPR) per International Myeloma Working Group (IMWG) criteria reported as proportion with 90% binomial confidence interval for the expansion cohort including the patients on MTD in the dose escalation cohort

SECONDARY OUTCOMES:
Duration of response | Up to 12 months following CAR- T infusion
  This is measured, only in responders, from the documented beginning of response (sCR, CR, PR or VGPR) to the time of progression per IMWG criteria for the expansion cohort including the patients on MTD in the dose escalation cohort
Progression-free Survival (PFS) | Up to 12 months following CAR- T infusion
  PFS is defined as the rate of survival from the the time from entry onto study until MM progression by IMWG criteria, or death from any cause for the expansion cohort including the patients on MTD in the dose escalation cohort.
Overall Survival | Up to 15 years
  Overall Survival is defined as the time from entry onto study until multiple myeloma progression or death from any cause. and will be be analyzed by Kaplan-Meier method for the expansion cohort including the patients on MTD in the dose escalation cohort.
Proportion of participants for whom BCMA CAR T-cell therapy is manufactured successfully | From initiation of CAR T-cell manufacturing to end of infusion, up to 21 days
  Participants who have anti-BCMA CAR T-cells successfully manufactured locally and are able to produce adequate quantities of vector positive T-cells which meet pre-specified release criteria.
Proportion of participants who complete study treatment | From initiation of CAR T-cell manufacturing to end of infusion, up to 21 days
  Participants who have anti-BCMA CAR T-cells successfully manufactured locally and are able to produce adequate quantities of vector positive T-cells which meet pre-specified release criteria which are then infused with the drug product.
Proportion of participants with treatment-emergent adverse events (AE) (Dose Expansion) | From initiation of CAR T-cell manufacturing to end of first follow-up, approximately 13 months
  Proportion of participants with treatment-emergent adverse events of CAR-T as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0, revised cytokine release syndrome CRS grading criteria (for CRS), and American Society of Transplantation and Cellular Therapy (ASTCT) Immune Effector Cell Associated Neurotoxicity (ICANS) Consensus Grading for Adults (for neurotoxicity).

CONTACTS AND LOCATIONS:
Overall Officials: Anupama Kumar, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No